CLINICAL TRIAL: NCT01318304
Title: Vaginal Innate Immunity in Normal and HIV-Infected Women
Status: Completed | Type: Observational
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Joseph Politch, Faculty, OBGYN, Boston Medical Center
Other Study IDs: H-29331
Record Dates: First submitted 2010-10-29; First posted 2011-03-18 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: HIV; Pregnancy
Keywords: innate immunity; HIV; pregnancy; vaginal immunity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Vaginal lavage samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Pregnant, HIV- negative: This cohort has completed accrual as of 12/28/11.
  Interventions: Other: Vaginal lavage specimen
- Pregnant, HIV-positive
  Interventions: Other: Vaginal lavage specimen
- Non-pregnant, HIV-negative: This cohort has completed accrual as of 12/28/11.
  Interventions: Other: Vaginal lavage specimen
- Non-pregnant, HIV-positive: This cohort has completed accrual as of 12/28/11.
  Interventions: Other: Vaginal lavage specimen

INTERVENTIONS:
Other: Vaginal lavage specimen — Collection of 3cc of saline used in the vagina to collect innate immunity markers

SUMMARY:
The innate immunity of the vaginal tract provides first-line defense from abnormal microorganisms or overgrowth of common organisms, such as Candida species or Gardnerella vaginalis. It is unclear from the current available literature whether the rate of vaginal infection increases or decreases in frequency during pregnancy when compared to the non-pregnant state, but this may be predicted by shifts in vaginal innate immunity. Vaginal infections are important players in HIV disease, potentially increasing the risk of viral transmission. In addition, these infections may activate inflammatory markers in the reproductive tract and increase the risk of premature delivery or other negative pregnancy outcomes. The vaginal innate immune system has not been well characterized in pregnant women, or in women with HIV infection. The study of how this system changes in pregnancy and HIV infection will provide essential knowledge for further study of vaginal mucosal protection.

The investigators study is an observational study designed to compare levels of vaginal innate immunity markers in women based on a) pregnancy status and b) HIV infection status. Comparisons will be made between pregnant and non- pregnant women and between HIV positive and HIV negative women. The investigators hypothesize that there will be significant differences in levels of innate immunity between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18 - 40 years
* Able to provide informed consent

Exclusion Criteria:

* Women with the following conditions will be excluded:
* Currently active Syphilis or Herpes simplex infection
* Other (non-HIV) comorbid conditions causing acute or chronic inflammatory states or immunosuppression (i.e., transplant recipients, active systemic lupus)
* Current use of hormonal birth control or with IUD in place
* History of Hysterectomy or bilateral oophorectomy

Women with the following conditions will require rescheduling of the study visit:

* Use of hot tub or pool, vaginal creams, douches, vaginal medications, or vaginal intercourse within 48 hours
* Current vaginal bleeding
* Recent treatment for vaginal infection will require 4 - 6 week delay in enrollment

Pregnant women with the following conditions at the time of examination will be excluded:

* Active labor or other conditions of duress
* Signs or symptoms of preterm labor
* Vaginal bleeding
* Placenta previa
* History of prior preterm birth
* Ruptured amniotic membranes
* Multifetal gestation
* Stillbirth or intrauterine fetal demise (IUFD)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy women, 18 to 40 years old, with spontaneous menstrual cycles or with normal ongoing pregnancy with gestational age between weeks 13 - 30 and able to provide informed consent
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2010-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
To compare the vaginal concentrations innate immunity markers (alpha / beta interferons, defensin, cathelicidin, lysozyme, lactoferrin, and SLPI) in pregnant and non-pregnant women who are HIV-negative. | up to 2 clinic visits in 10 weeks
  Investigators will quantify the major vaginal innate immunity markers, including type 1 (alpha and beta) interferons, defensins, cathelicidins, lysozyme and lactoferrin, and secretory leukocyte protease inhibitor (SLPI). These antimicrobial host defense peptides are produced by genital tract mucosal epithelial cells and associated immune cells, and have a wide range of antiviral, antibacterial, antifungal and antiparasitic activities and modes of action. We hypothesize that changes in innate immunity markers take place during pregnancy, thereby changing native vaginal immunity.

SECONDARY OUTCOMES:
To compare the vaginal concentrations of innate immunity markers (alpha and beta) interferon, defensin, cathelicidin, lysozyme, lactoferrin, and SLPI)) in HIV-positive pregnant and non-pregnant women | up to 2 clinic visits in 10 weeks
  Investigators will quantify the major vaginal innate immunity markers, including type 1 (alpha and beta) interferons, defensins, cathelicidins, lysozyme and lactoferrin, and secretory leukocyte protease inhibitor (SLPI). Women who have HIV may express different innate immunity marker profiles in vaginal secretions when pregnant as compared to non-pregnant HIV positive women. Timing of specimen collection: In pregnancy: Weeks 13 - 30. Non-pregnant: 3 weeks between menstrual bleeding cycles
To compare the vaginal concentrations innate immunity markers (alpha / beta interferons, defensin, cathelicidin, lysozyme, lactoferrin, and SLPI) in pregnant women who are HIV-negative to pregnant women who are HIV-positive. | up to 2 clinic visits in 10 weeks
  Investigators will quantify the major vaginal innate immunity markers, including type 1 (alpha and beta) interferons, defensins, cathelicidins, lysozyme and lactoferrin, and secretory leukocyte protease inhibitor (SLPI). Women with HIV may express different innate immunity marker profiles in vaginal secretions when pregnant as compared to pregnant, HIV-negative women. This may provide some explanation for differences in vaginal infection rates between the groups. Timing of specimen collection: In pregnancy: Weeks 13 - 30.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Ballard Dwan, M.D., Principal Investigator — Boston University; Deborah Anderson, Ph.D., Principal Investigator — Boston University
Locations (1):
- Boston University Medical Center, Boston, Massachusetts, United States